CLINICAL TRIAL: NCT01135004
Title: Molecular Pathogenesis of Primary Spontaneous Pneumothorax
Brief Title: Pathogenesis of Primary Spontaneous Pneumothorax
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Yung-Chie Lee, Professor, National Taiwan University Hospital
Other Study IDs: 200912060R
Record Dates: First submitted 2010-05-30; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-03

CONDITIONS: Pneumothorax
Keywords: pneumothorax; thoracoscopy; pathogenesis; blebs; surgery
MeSH Terms: conditions — Pneumothorax; Blister | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Thoracoscopic bullectomy will be performed in spontaneous pneumothorax patients. Part of the surgcal specimen (lung tissue) will be obtained for RNA and protein analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pneumothorax patients: Primary spontaneous pneumothorax patients undergoing thoracoscopic bullectomy
  Interventions: Procedure: Thoracoscopic bullectomy

INTERVENTIONS:
Procedure: Thoracoscopic bullectomy — Thoracoscopic wedge resection of the diseased lung
  Other Names: Video-assisted thoracic surgery (VATS)

SUMMARY:
Primary spontaneous pneumothorax most commonly occurs in young, tall, lean males. The estimated recurrence rate is 23-50% after the first episode and increases to 60% after the second pneumothorax. The pathogenesis of this benign disease remains unclear. Generally, rupture of the emphysematous change or blebs in the apex of the lung is considered as the cause of pneumothorax. The main purpose of this study is to investigate the molecular pathogenesis of blebs formation or emphysematous change of the lung in these young, healthy patients.

DETAILED DESCRIPTION:
Primary spontaneous pneumothorax most commonly occurs in young, tall, lean males. The estimated recurrence rate is 23-50% after the first episode and increases to 60% after the second pneumothorax. The pathogenesis of this benign disease remains unclear. Generally, rupture of the emphysematous change or blebs in the apex of the lung is considered as the cause of pneumothorax. The main purpose of this study is to investigate the molecular pathogenesis of blebs formation or emphysematous change of the lung in these young, healthy patients. The blebs resected from the pneumothorax patients will be used for RNA and protein levels analyses. The adjacent normal lung tissue will be used as a control for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 and 40 years
* Spontaneous pneumothorax
* Underwent bullectomy of the lung

Exclusion Criteria:

* With underlying lung disease

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary spontaneous pneumothorax most commonly occurs in young, tall, lean males without underlying pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-02 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Ayed AK, Chandrasekaran C, Sukumar M. Video-assisted thoracoscopic surgery for primary spontaneous pneumothorax: clinicopathological correlation. Eur J Cardiothorac Surg. 2006 Feb;29(2):221-5. doi: 10.1016/j.ejcts.2005.11.005. Epub 2005 Dec 20. PMID 16376095